CLINICAL TRIAL: NCT06521866
Title: A Prospective, Randomized, Phase II, Multicenter Clinical Study of Serplulimab Combined with First-Line Targeted Therapy and Chemotherapy with or Without Radiation in the First-Line Treatment of Advanced Colorectal Cancer
Brief Title: Phase II Study of Serplulimab Combined with First-Line Targeted Therapy, Chemotherapy, and Radiation in Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Li Dawei, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICTORY CRC
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Advanced Colorectal Carcinoma; Immunotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Experimental): Group A (Left-sided wild-type):
  Induction Treatment (12 cycles):
  Serplulimab: IV 3 mg/kg on Day 1, q2w Cetuximab: 400 mg/m² IV infusion (1st infusion >2 hours, then 250 mg/m² IV infusion ≥60 min), weekly mFOLFOX6: Oxaliplatin: 85 mg/m² IV over 2 hrs, Day 1 LV: 400 mg/m² IV over 2 hrs, Day 1 5-FU: 400 mg/m² IV push, Day 1; 2400 mg/m² IV over 46-48 hrs q2w
  Maintenance therapy:
  Serplulimab: IV 3 mg/kg on Day 1, q2w Cetuximab: 400 mg/m² IV infusion (1st infusion >2 hours, then 250 mg/m² IV infusion ≥60 min), weekly 5-FU/LV: LV: 400 mg/m² IV over 2 hrs, Day 1 5-FU: 400 mg/m² IV push, Day 1; 2400 mg/m² IV over 46-48 hrs q2w
  Interventions: Drug: Serplulimab; Drug: Chemotherapy; Drug: Targeted therapy
- Group B (Experimental): Group B (Left-sided wild-type):
  One cycle of Serplulimab combined with Cetuximab and chemotherapy, followed by Stereotactic ablative radiotherapy（SABR: 25-60 Gy/5 Fx）, then continued Serplulimab combined with Cetuximab and chemotherapy.
  Interventions: Drug: Serplulimab; Drug: Chemotherapy; Radiation: SABR; Drug: Targeted therapy
- Group C (Experimental): Group C (Right-sided or RAS-mutant): Induction Treatment (12 cycles):
  Serplulimab: IV 3 mg/kg on Day 1, q2w Bevacizumab: 5 mg/kg IV on Day 1, q2w mFOLFOX6: Oxaliplatin: 85 mg/m² IV over 2 hrs, Day 1 LV: 400 mg/m² IV over 2 hrs, Day 1 5-FU: 400 mg/m² IV push, Day 1; 2400 mg/m² IV over 46-48 hrs q2w
  Maintenance Treatment:
  Serplulimab: IV 3 mg/kg on Day 1, q2w Bevacizumab: 5 mg/kg IV on Day 1, q2w 5-FU/LV: LV: 400 mg/m² IV over 2 hrs, Day 1 5-FU: 400 mg/m² IV push, Day 1; 2400 mg/m² IV over 46-48 hrs q2w
  Interventions: Drug: Serplulimab; Drug: Chemotherapy; Drug: Targeted therapy
- Group D (Experimental): Group D (Right-sided or RAS-mutant): One cycle of Serplulimab combined with Bevacizumab and chemotherapy, followed by Stereotactic ablative radiotherapy（SABR: 25-60 Gy/5 Fx）, then continued Serplulimab combined with Bevacizumab and chemotherapy.
  Interventions: Drug: Serplulimab; Drug: Chemotherapy; Radiation: SABR; Drug: Targeted therapy

INTERVENTIONS:
Drug: Serplulimab — IV 3 mg/kg on Day 1, q2w
Drug: Chemotherapy — Induction therapy：Oxaliplatin: 85 mg/m² IV on Day 1 Leucovorin (LV): 400 mg/m² IV on Day 1 5-FU: 400 mg/m² IV bolus on Day 1, then 2400 mg/m² continuous IV infusion over 46-48 hours
  Maintenance therapy:
  Leucovorin (LV): 400 mg/m² IV on Day 1 5-FU: 400 mg/m² IV bolus on Day 1, then 2400 mg/m² continuous IV infusion over 46-48 hours
Radiation: SABR — SABR: 25-60 Gy/5 Fx
  Arms: Group B; Group D
Drug: Targeted therapy — Cetuximab: 400 mg/m² IV on Day 1, then 250 mg/m² IV weekly ; Bevacizumab: 5 mg/kg IV on Day 1

SUMMARY:
Study Title:

A Prospective, Randomized, Phase II, Multicenter Clinical Study of Serplulimab Combined with Targeted Therapy, Chemotherapy, and Optional Radiotherapy in Advanced Colorectal Cancer

Study Objective:

To explore the efficacy and safety of immune checkpoint inhibitor combined with targeted therapy and chemoradiotherapy in locally advanced unresectable or metastatic colorectal cancer.

Study Population:

Patients with left-sided wild-type, right-sided, or RAS-mutant advanced colorectal cancer who have not received systemic treatment.

Study Endpoints:

Progression-free survival (PFS), objective response rate (ORR), overall survival (OS), safety, and R0 resection rate.

Study Design:

Prospective, randomized Phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, any gender;
2. Histologically confirmed metastatic colorectal cancer (Stage IV, UICC), with initially unresectable metastases or refusal of surgery;

   * Primary tumor located in the distal transverse colon, descending colon, sigmoid colon, and rectum, and RAS (KRAS and NRAS) and BRAF wild-type (Cohorts A and B);
   * Primary tumor located in the cecum, ascending colon, and proximal transverse colon, and RAS (KRAS and NRAS) mutant-type (Cohorts C and D);
3. Treatment-naive patients who have not received standard anti-tumor therapy;
4. At least one measurable tumor lesion per RECIST 1.1 criteria;
5. ECOG performance status of 0-1;
6. Patients with an expected survival time of ≥ 3 months and good organ function:

   * (1) Neutrophils ≥ 1.5 * 10^9/L; platelets ≥ 100 * 10^9/L; hemoglobin ≥ 9 g/dL; serum albumin ≥ 3 g/dL;
   * (2) Thyroid-stimulating hormone (TSH) ≤ upper limit of normal (ULN), T3 and T4 within normal ranges;
   * (3) Bilirubin ≤ 1.5 times ULN; ALT and AST ≤ 2 times ULN;
   * (4) Serum creatinine ≤ 1.5 times ULN, creatinine clearance rate ≥ 60 mL/min;
   * (5) International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN, unless the patient is receiving anticoagulant therapy and PT is within the expected therapeutic range of anticoagulants;
   * (6) Activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN;
7. Female patients of childbearing potential must have a negative pregnancy test; female patients not of childbearing potential; male patients of reproductive potential and female patients of reproductive potential and at risk of pregnancy must agree to use adequate contraception throughout the study period, continuing until 12 months after the last dose of study treatment;
8. Signed and dated informed consent form indicating that the patient has been informed of all pertinent aspects of the study;
9. Patients willing and able to comply with visit schedule, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Pathologically diagnosed with other intestinal tumors, such as gastrointestinal stromal tumors;
2. No testing for RAS mutation status;
3. Resectable metastases or patients wishing to undergo metastasectomy;
4. Prior systemic therapy. Systemic therapy includes all of the following: chemotherapy agents such as fluoropyrimidines, irinotecan, and oxaliplatin, VEGF monoclonal antibodies (e.g., bevacizumab), EGFR monoclonal antibodies (cetuximab or panitumumab), small molecule TKIs, immune checkpoint inhibitors, etc.;
5. Uncontrolled active bleeding from the primary tumor or bowel obstruction;
6. Contraindications to immune checkpoint inhibitors;
7. Allergy to the therapeutic drugs and/or their excipients;
8. Previous treatment with PD-1 antibodies, PD-L1 antibodies, or CTLA-4 antibodies;
9. Received any form of radiation therapy within 4 weeks prior to enrollment;
10. Previous or concurrent other malignancies, except adequately treated non-melanoma skin cancer, in situ cervical cancer, or papillary thyroid carcinoma;
11. Active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); except autoimmune-mediated hypothyroidism on stable doses of thyroid replacement hormone, type I diabetes on stable doses of insulin, vitiligo, or childhood asthma/allergies that have resolved and do not require intervention in adulthood;
12. History of immunodeficiency, including HIV-positive, or other acquired/congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation;
13. History of interstitial lung disease (excluding radiation pneumonitis not treated with steroids), non-infectious pneumonia;
14. Active tuberculosis infection identified by history or CT scan, or history of active tuberculosis infection within 1 year prior to enrollment, or history of active tuberculosis infection more than 1 year ago but without proper treatment;
15. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL), active hepatitis C (HCV antibody positive and HCV-RNA above the detection limit);
16. Severe dysfunction of the heart, lungs, or kidneys;
17. Hypertension not well controlled by antihypertensive medications (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
18. History of substance abuse, alcoholism, or drug addiction;
19. Any other factors judged by the investigator to potentially affect the safety or compliance of the patient with the study, such as serious concomitant disease (including mental illness), serious laboratory abnormalities, or other familial or social factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 year
  Progression Free Survival

SECONDARY OUTCOMES:
OS | 2 year
  Overall Survial
ORR | 2 year
  Objective Response Rate
Incidence of Side Effect | 2 year
  Side Effect

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou Military Region General Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huai'an Second People's Hospital, Huaian, Jiangsu
  - Qianfoshan Hospital of Shandong Province, Jinan, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Anyang Cancer Hospital, Anyang

IPD SHARING:
Plan to Share IPD: Undecided